CLINICAL TRIAL: NCT06120218
Title: Tandem Occlusion After Emergent Stenting in Acute Ischemic Stroke: Preliminary Experience From a Vietnamese Comprehensive Stroke Centre
Brief Title: Tandem Occlusion After Emergent Stenting in Acute Ischemic Stroke
Acronym: TOESIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho Stroke International Services Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cuong Tran Chi, Director, Can Tho Stroke International Services Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOESIS Study
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Acute Stroke; Ischemic Stroke, Acute
Keywords: Thrombectomy; Extracranial arteries; Endovascular treatment; Antegrade approach; Retrograde approach
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergent Stenting in Anterior circulation (Experimental): Emergent Carotid Stenting in acute ischemic stroke caused by tandem occlusions
  Interventions: Procedure: Emergent Stenting
- Emergent Stenting in Posterior circulation (Experimental): Emergent Extracranial Vertebral Stenting in acute ischemic stroke caused by tandem occlusions
  Interventions: Procedure: Emergent Stenting

INTERVENTIONS:
Procedure: Emergent Stenting — Emergent Stenting in acute ischemic stroke caused by tandem occlusions

SUMMARY:
In acute ischemic stroke due to tandem occlusion, the emergent stenting has recently become an endovascular treatment option combining with mechanical thrombectomy to achieve recanalization. However, the data on the beneficial endovascular management of tandem occlusion in two circulations is still limited. The purpose of our study was to compare the improvement of clinical outcome between two circulations after emergent stenting at 3 months.

DETAILED DESCRIPTION:
The posterior circulation (about 20 - 25%) is less frequent than the anterior one in the acute ischemic stroke, but high mortality and morbidity in the acute vertebrobasilar thrombosis even successful recanalization are revealed. Besides, tandem occlusion is one of the complex lesions in large vessel occlusions relating to the poor outcome, particularly in the posterior circulation. Recent studies have suggested that emergent stenting could be used as an additional treatment to achieve permanent recanalization together with mechanical thrombectomy in the intracranial segments. Permanent recanalization is one of the most important factors that impact patient outcomes after acute ischemic stroke. However, although there are various approaches for this lesion, the comparision of the effectiveness in the two circulations remains unclear. Thus, the aims of our study were to compare baseline characteristics and clinical outcome of tandem occlusions between anterior and posterior circulation after emergent stenting in extracranial arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Premorbid mRS < 2
* NIHSS > 5
* ASPECTS ≥ 5 or pc-ASPECTS ≥ 5

Exclusion Criteria:

* Onset to treatment time > 24 hours
* Loss to follow up after discharge

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The favorable 3-month outcome rate | 3 months
  The favorable 3-month outcome rate was accessed by modified Rankin Score (mRS), which comprised of included good (mRS 0 - ≤ 2) and fair (mRS 3).

SECONDARY OUTCOMES:
The symptomatic intracerebral hemorrhage rate | 24 hours after emergent stenting
  The symptomatic intracerebral hemorrhage was defined as patient's intracerebral hemorrhage with postprocedural mRS ≥ 5 and there were no other evident causes for the increased modified Rankin Score (mRS).

CONTACTS AND LOCATIONS:
Overall Officials: Cuong Tran Chi, Doctor, Study Director — Can Tho Stroke International Services General Hospital
Locations (1):
- Can Tho Stroke International Services Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allard J, Delvoye F, Pop R, Labreuche J, Maier B, Marnat G, Sibon I, Zhu F, Lapergue B, Consoli A, Spelle L, Denier C, Richard S, Piotin M, Gory B, Mazighi M; ETIS Investigators. 24-Hour Carotid Stent Patency and Outcomes After Endovascular Therapy: A Multicenter Study. Stroke. 2023 Jan;54(1):124-131. doi: 10.1161/STROKEAHA.122.039797. Epub 2022 Dec 21. PMID 36542074
- [Background] Han N, Ma L, Zhao L, Xu G, Jia Y, Wang H. The Dilator-Dotter technique can successfully treat tandem lesions of posterior circulation. Medicine (Baltimore). 2024 Jan 26;103(4):e37044. doi: 10.1097/MD.0000000000037044. PMID 38277540